CLINICAL TRIAL: NCT01556802
Title: Effect of Minocicline Use in Less Neurologic Sequels in Patients With Stroke
Brief Title: Use of Minocicline in Patients With Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Hernando Moncaleano Perdomo (Other)
Responsible Party: Principal Investigator, Nataly Bedoya, Internist, Hospital Universitario Hernando Moncaleano Perdomo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 38212050
Record Dates: First submitted 2012-03-05; First posted 2012-03-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Stroke; Brain Ischemia; Paralysis
Keywords: stroke; sequelaes; minocicline
MeSH Terms: conditions — Stroke; Brain Ischemia; Paralysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocicline (Experimental): minocicline 100mg oral twice a day for 5 days
  Interventions: Drug: Minocicline
- Placebo (Placebo Comparator): Pills filled with vegetal fiber with similar presentation of the drug. Given one pill oral twice a day for five days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocicline — Minocicline 100mg oral twice a day for 5 days
  Arms: Minocicline
Drug: Placebo — Pills with vegetable fibers one pill oral twice a day for five days
  Arms: Placebo

SUMMARY:
The investigators will evaluate the National Institute of Health Stroke Scale/Score (NIHSS)in patients with stroke, and then give Minocycline 100mg po every 12 hours or placebo for five days, then perform periodic evaluations to determine the status and degree of neurological sequelae developed.

ELIGIBILITY:
Inclusion Criteria:

* NIHSS scale greater than 5
* Onset of symptoms less than 24 hours
* normal Cranial Tomography(CT)
* CT evidence of cerebral ischemia
* Acceptance of study entry

Exclusion Criteria:

* Hemorrhagic cerebrovascular disease
* Other neurological diseases
* Concomitant structural damage
* History of neurosurgery
* Known allergy to tetracyclines
* Concomitant infectious diseases requiring antibiotic treatment.
* History of Stroke
* Women pregnant or breast-feeding

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of minocycline in reducing neurological sequelae in patients with stroke | one year
  The researchers evaluated the neurological condition of paralysis, aphasia,and level of consciousness by NIHSS score for each patient with stroke and proceeded to give minocycline or placebo. Then, the assessment was repeated after five and thirty days post treatment to determine whether their neurological sequelae had diminushed.

SECONDARY OUTCOMES:
Identify the side effects of the intervention administered during the treatment time and 30 days later. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nataly Bedoya, Internist, Study Director — Universidad Surcolombiana; Hernan Vargas, Internist, Principal Investigator — Universidad Surcolombiana; Hugo Osorio, Internist, Principal Investigator — Universidad Surcolombiana; Guillermo Gonzalez, Neurologist, Principal Investigator — Universidad Surcolombiana; Javier Saldaña, Epidemiology, Principal Investigator — Universidad Surcolombiana; Efrain Amaya, Neurologist, Principal Investigator — Hospital Hernando Moncaleano Perdomo
Locations (1):
- University Hospital hernando Moncaleano Perdomo, Neiva, Huila Department, Colombia